CLINICAL TRIAL: NCT00749463
Title: Evaluation of the Safety Profile, Quit and Reduction Rate After Nicorette® Gum and Patch Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP4009
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: nicotine dependence, smoking cessation, NRT
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gum 2 (Experimental): Nicotine Gum 2 mg for subjects smoking less than 20 cigarettes per day; 2 mg for 12 week treatments and followed by 12 week off-treatment follow-up. Recommend subject to use 8-12 pieces daily for first 8 weeks and 4-6 pieces daily the next 2 weeks, then reduce to 1-3 pieces each day in last 2 weeks
  Interventions: Drug: Nicotine Gum
- Gum 4 (Experimental): Nicotine Gum 4 mg for subjects smoking 20 or more cigarettes per day; 4 mg for 12 week treatments and followed by 12 week off-treatment follow-up. Recommend subject to use 8-12 pieces daily for first 8 weeks and 4-6 pieces daily the next 2 weeks, then reduce to 1-3 pieces each day in last 2 weeks
  Interventions: Drug: Nicotine Gum
- Patch (Experimental): Nicotine Patch; Each will use 15 mg/16 h patch for the first 8 weeks, 10 mg/16 h for the following 2 weeks and 5 mg/16 h for the last 2 weeks. Then followed by 12 week off-treatment follow-up.
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Drug: Nicotine Gum — 2 mg or 4 mg for 12 week treatments and followed by 12 week off-treatment follow-up. Recommend subject to use 8-12 pieces daily for first 8 weeks and 4-6 pieces daily the next 2 weeks, then reduce to 1-3 pieces each day in last 2 weeks
  Other Names: Nicorette® Gum
  Arms: Gum 2; Gum 4
Drug: Nicotine Patch — Each will use 15 mg/16 h patch for the first 8 weeks, 10 mg/16 h for the following 2 weeks and 5 mg/16 h for the last 2 weeks. Then followed by 12 week off-treatment follow-up.
  Other Names: Nicorette® Patch
  Arms: Patch

SUMMARY:
To evaluate the safety, smoking cessation and reduction rate during 3 months of active nicotine replacement therapy (NRT) and a follow-up period of 3 months in smoking hospital physicians and staff who are motivated to quit

DETAILED DESCRIPTION:
Using Nicorette® gum 2 mg, 4 mg and Nicorette® patch 5 mg/16 h, 10 mg/16 h, 15 mg/16 h to alleviate nicotine cravings and withdrawal symptoms and assist smoking cessation in smoking hospital physicians and staff who are motivated to quit. During the study, brief telephone consultation and SMS are provided as behavioral supports.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, aged 18 years or older
* Normal dental status and chewing ability for nicotine gum users; normal skin without excessive hair growth on tested areas for nicotine patch users
* Current daily smoker for at least two years
* Have a carbon monoxide (CO) level of at least 10 parts per million (ppm) after at least 15 smoke-free minutes
* Be motivated to stop smoking with the help of nicotine gum or patch treatment.
* Evidence of a personally signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the trial
* Be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Current use of other tobacco-containing products e.g. snuff, chewing tobacco, cigars, or pipes.
* Use of any other stop-smoking products (nicotine or non-nicotine) or treatment (hypnosis, acupuncture, etc) during the study i.e. during the last 6-month period.
* Unstable angina pectoris or myocardial infarction during the previous 3 months.
* Pregnancy, lactation or intended pregnancy.
* Any major metabolic disease, clinically important renal, hepatic disease.
* Suspected alcohol or drug abuse.
* Participation in other clinical trials in the previous three months, or during study participation.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Mao, Study Chair — Shanghai Johnson & Johnson Pharmaceuticals
Locations (6):
- China (6):
  - Beijing ChaoYang Hospital, Beijing, Beijing Municipality
  - People's Hospital affiliated to Beijing University, Beijing, Beijing Municipality
  - No. 1 Hospital affiliated to Zhongshan University, Guangzhou, Guangdong
  - No. 1 Hospital affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Chang Zheng Hospital, Shanghai, Shanghai Municipality
  - Zhong Shan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Gum 2: Dosage: 2 mg, Dosage Form: Gum
- Nicotine Gum 4: Dosage: 4 mg, Dosage Form: Gum
- Nicotine Patch: Dosage: Step-down treatment 15 mg,10 mg, then 5 mg/16 hours Dosage Form: Patch
Period: Overall Study
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Started | 86 | 64 | 150
Completed | 85 | 60 | 149
Not Completed | 1 | 4 | 1
Not completed — Adverse Event | 0 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch | Total
Number analyzed (Participants) | 86 | 64 | 150 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.2) | 40.3 (10.0) | 41.7 (11.6) | 41.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 86 | 62 | 149 | 297
Region of Enrollment [Number; unit: participants]
  China | 86 | 64 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Related Adverse Events
Description: Percentage of subjects with treatment-related adverse events by preferred term, included if the percentage in any single arm was 1% or higher
Time Frame: 24 Weeks
Population: Safety Analysis Set (ITT)
Measure: Number; unit: Percentage of Participants
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 86 | 64 | 150
Percentage of Participants
  Subjects with at Least One Treatment-Related AE | 25.6 | 39.1 | 21.3
  Sinus tachycardia | 0 | 1.6 | 0
  Abdominal distension | 2.3 | 0 | 0
  Abdominal pain upper | 3.5 | 1.6 | 0.6
  Abdominal symptom | 1.2 | 0 | 0
  Diarrhoea | 0 | 1.6 | 0.6
  Dyspepsia | 1.2 | 1.6 | 0
  Eructation | 0 | 1.6 | 0
  Gingival ulceration | 0 | 1.6 | 0
  Mouth ulceration | 2.3 | 0 | 0.6
  Nausea | 15.1 | 21.9 | 5.3
  Oral discomfort | 1.2 | 0 | 0
  Retching | 0 | 1.6 | 0
  Chest discomfort | 1.2 | 3.1 | 0
  Heart rate increased | 0 | 1.6 | 0
  Myalgia | 0 | 1.6 | 0
  Dizziness | 1.2 | 1.6 | 2.0
  Insomnia | 0 | 0 | 1.3
  Hiccups | 0 | 1.6 | 0
  Oropharyngeal pain | 8.1 | 7.8 | 0.6
  Tachypnoea | 1.2 | 1.6 | 0
  Dermatitis allergic | 0 | 0 | 8.0
  Pruritus | 0 | 0 | 2.0
  Rash vesicular | 0 | 0 | 1.3

2. Primary Outcome: Self-Reported Smoking Reduction
Description: Percentage of subjects self-reporting reduction from baseline in number of cigarettes smoked per day
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 86 | 64 | 150
Percentage of Participants
  Week 1 | 78.8 (24.3) | 73.6 (21.9) | 75.2 (25.1)
  Week 2 | 79.9 (22.0) | 73.5 (21.6) | 77.0 (24.4)
  Week 3 | 81.0 (22.6) | 77.3 (22.2) | 79.9 (23.7)
  Week 4 | 84.2 (20.1) | 78.6 (23.6) | 80.3 (24.2)
  Week 6 | 81.0 (23.6) | 78.0 (22.8) | 77.2 (26.7)
  Week 8 | 80.8 (23.5) | 75.4 (24.6) | 77.1 (28.9)
  Week 10 | 80.9 (24.5) | 76.0 (24.0) | 77.6 (27.7)
  Week 12 | 80.8 (24.1) | 77.0 (22.0) | 78.7 (27.5)
  Week 16 | 76.0 (27.1) | 72.3 (26.3) | 74.8 (31.6)
  Week 20 | 73.7 (29.7) | 69.3 (28.5) | 74.0 (32.6)
  Week 24 | 72.7 (31.6) | 63.7 (31.0) | 71.9 (34.0)

3. Secondary Outcome: Carbon Monoxide (CO)-Verified Smoking Reduction
Description: Percentage of participants with carbon monoxide (CO)-verified reduction from baseline in number of cigarettes smoked per day (%)
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 86 | 64 | 150
Percentage of Participants
  Visit at 2 Weeks | 82.3 (21.1) | 76.1 (20.0) | 80.6 (19.0)
  Visit at 6 Weeks | 83.7 (20.4) | 78.9 (22.4) | 81.6 (21.0)
  Visit at 8 Weeks | 86.1 (18.0) | 77.4 (23.4) | 81.9 (23.3)
  Visit at 10 Weeks | 85.1 (18.9) | 78.7 (20.0) | 82.9 (22.2)
  Visit at 12 Weeks | 84.7 (19.4) | 79.5 (19.8) | 83.4 (23.6)
  Visit at 24 Weeks | 80.4 (25.5) | 67.6 (29.2) | 81.2 (25.5)

4. Secondary Outcome: Smoking Consumption Per Day
Description: Number of cigarettes smoked by subjects reporting smoking since last visit - total during the day (for daily smokers)
Time Frame: 24 Weeks from last visit:
Measure: Mean (Standard Deviation); unit: Cigarettes
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 35 | 37 | 67
Cigarettes | 9.5 (6.3) | 16.1 (8.2) | 11.9 (8.2)

5. Secondary Outcome: Smoking Consumption Per Week
Description: Number of cigarettes smoked by subjects reporting smoking since last visit - total during the the week (for non-daily smokers)
Time Frame: 24 Weeks from last visit:
Measure: Mean (Standard Deviation); unit: Cigarettes
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 18 | 7 | 25
Cigarettes | 25.8 (21.4) | 41.6 (27.7) | 22.1 (24.6)

6. Primary Outcome: Smoking Abstinence
Description: Continuous carbon monoxide (CO)-verified Smoking Abstinence from Quit day
Time Frame: 24 Weeks
Measure: Number; unit: Participants
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 86 | 64 | 150
Participants
  Visit at 2 Weeks | 24 | 9 | 34
  Visit at 6 Weeks | 19 | 7 | 24
  Visit at 8 Weeks | 18 | 7 | 24
  Visit at 10 Weeks | 17 | 7 | 22
  Visit at 12 Weeks | 16 | 7 | 21
  Visit at 24 Weeks | 13 | 7 | 17

7. Secondary Outcome: Point Prevalence Smoking Abstinence (PPSA)
Description: Point Prevalence Smoking Abstinence since last visit. Point prevalence abstinence is defined as the percentage of former smokers who are not smoking at a particular point in time, typically at the time of assessment.
Time Frame: 24 Weeks
Measure: Number; unit: Participants
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Number analyzed (Participants) | 86 | 64 | 150
Participants
  Week 1 | 28 | 11 | 42
  Week 2 | 28 | 13 | 43
  Week 3 | 33 | 15 | 50
  Week 4 | 33 | 16 | 55
  Week 6 | 31 | 16 | 45
  Week 8 | 33 | 16 | 50
  Week 10 | 32 | 16 | 51
  Week 12 | 34 | 16 | 60
  Week 16 | 33 | 17 | 53
  Week 20 | 32 | 17 | 55
  Week 24 | 32 | 16 | 57

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Nicotine Gum 2 | Nicotine Gum 4 | Nicotine Patch
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/64 | 0/150
Other Adverse Events (participants affected / at risk) | 22/86 | 26/64 | 33/150
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Gum 2 (N=86) | Nicotine Gum 4 (N=64) | Nicotine Patch (N=150)
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal symptom (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 15 | 8
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 2 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less